CLINICAL TRIAL: NCT00104975
Title: Reduced Intensity Conditioning Regimen for Haplo-identical Family Donor Stem Cell Transplants for Hematologic Malignancies With Delayed Add-back of Non-alloreactive T Cells
Brief Title: Alemtuzumab and Combination Chemotherapy Followed By Donor Lymphocytes in Treating Patients Who Are Undergoing Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000413698; YALE-25971; NCI-6765
Record Dates: First submitted 2005-03-03; First posted 2005-03-04 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms
Keywords: accelerated phase chronic myelogenous leukemia; recurrent adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; recurrent adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; refractory anemia with excess blasts in transformation; refractory anemia with excess blasts; secondary myelodysplastic syndromes; chronic myelomonocytic leukemia; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; refractory chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; stage III adult Burkitt lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; myelodysplastic/myeloproliferative neoplasm, unclassifiable; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Leukemia, Myeloid, Accelerated Phase; Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Large-Cell, Immunoblastic; Anemia, Refractory, with Excess of Blasts; Leukemia, Myelomonocytic, Chronic; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — Alemtuzumab; fludarabine phosphate; Melphalan; Tacrolimus; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: alemtuzumab
Biological: therapeutic allogeneic lymphocytes
Drug: fludarabine phosphate
Drug: melphalan
Drug: tacrolimus
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Giving low doses of chemotherapy before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune system and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells that have been treated in the laboratory after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus before and after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of donor lymphocytes when given after alemtuzumab and combination chemotherapy in treating patients who are undergoing donor stem cell transplant for hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and efficacy of a reduced-intensity conditioning regimen comprising alemtuzumab, fludarabine, melphalan, and thiotepa followed by allogeneic peripheral blood stem cell transplantation (PBSCT) in patients with hematologic malignancies.
* Determine the toxicity of this regimen in these patients.
* Determine the safety of LMB-2 immunotoxin-treated, selectively-depleted donor T cells, administered after allogeneic PBSCT, in these patients.

OUTLINE: This is a dose-escalation study of LMB-2 immunotoxin-treated, selectively-depleted donor T cells.

* T cell preparation: Patients and donors undergo apheresis to obtain peripheral blood mononuclear cells (PBMCs), which are expanded in culture. Patients' PBMCs are irradiated and mixed with donor PBMCs. LMB-2 immunotoxin is added to the PBMCs in order to selectively deplete T cells from the donor PBMCs.
* Conditioning: Patients receive alemtuzumab IV over 2 hours on days -9 to -5, fludarabine IV over 30 minutes on days -8 to -5, melphalan IV over 15-20 minutes on day -4, and thiotepa IV on days -3 to -2.
* Immunosuppression: Patients receive tacrolimus IV continuously on days -10 to 1.
* Allogeneic peripheral blood stem cell (PBSC) transplantation: Patients undergo allogeneic PBSC transplantation on day 0.
* LMB-2 immunotoxin-treated, selectively-depleted donor T cells: Patients receive LMB-2 immunotoxin-treated, selectively-depleted donor T cells IV over 30-60 minutes on approximately day 28.

Cohorts of 3-6 patients receive escalating dose of LMB-2 immunotoxin-treated, selectively-depleted donor T cells until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting-toxicity.

After completion of study treatment, patients are followed weekly for 100 days post-transplantation and then periodically for survival.

PROJECTED ACCRUAL: A total of 15-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic malignancies:

  * Chronic myelogenous leukemia

    * Accelerated phase or blast phase
  * Acute myeloid leukemia, meeting any of the following criteria:

    * In second or subsequent remission
    * In primary induction failure
    * In partial remission
    * In resistant relapse
  * Chronic lymphocytic leukemia

    * In Richter's transformation
  * High-grade non-Hodgkin's lymphoma

    * Refractory to standard treatment
  * Myeloproliferative disorders

    * Undergoing transformation to terminal stages
  * Myelodysplastic syndromes (MDS), including any of the following:

    * Refractory anemia with excess blasts
    * Transformation to acute leukemia
    * MDS secondary to chemotherapy
* Partially-matched related family donor available

  * One HLA haplotype match
* No HLA-matched (10/10 or 9/10) sibling donor or unrelated donor available NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age

* 18 to 55

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* SGOT and SGPT < 3 times upper limit of normal (ULN)
* No active or persistent viral hepatitis

Renal

* Creatinine < 2.0 mg/dL* OR
* Creatinine clearance > 60 mL/min* NOTE: *Unless due to malignancy

Cardiovascular

* LVEF ≥ 45%

Pulmonary

* DLCO ≥ 60% of predicted* (corrected for hemoglobin) NOTE: *Unless patient is given clearance by a pulmonary consultation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for up to 2 years after completion of study treatment
* HIV negative
* Human T cell lymphotrophic virus type 1 negative
* No serious co-morbid medical condition
* No other medical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-02; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erkut Bahceci, MD, Study Chair — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States